CLINICAL TRIAL: NCT02547792
Title: Phase 1 , Placebo-Controlled, Dose-Ranging Trial to Determine Safety and Immunogenicity of an Oral Adenoviral-Vector Based Influenza B Vaccine
Brief Title: Assessment of an Oral Influenza B Vaccine Tablet (VXA-BYW.10) Following Single Dose Administration in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VXA03-001
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Seasonal Influenza B
Keywords: Influenza B
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VXA-BYW.10 (Low Dose) Oral Vaccine (Experimental): Single administration of Influenza B (Low Dose) oral vaccine tablets
  Interventions: Biological: VXA-BYW.10 (Low Dose) Oral Vaccine
- VXA-BYW.10 (High Dose) Oral Vaccine (Experimental): Single administration of Influenza B (High Dose) oral vaccine tablets
  Interventions: Biological: VXA-BYW.10 (High Dose) Oral Vaccine
- Placebo Tablets (Placebo Comparator): Matching placebo dose (size and number of tablets) to low dose vaccine (part 1) and high dose (part 2)
  Interventions: Other: Placebo Tablets

INTERVENTIONS:
Biological: VXA-BYW.10 (Low Dose) Oral Vaccine — Enteric coated tablet for oral delivery
  Other Names: Influenza B (Low Dose) Oral Vaccine Tablets
  Arms: VXA-BYW.10 (Low Dose) Oral Vaccine
Biological: VXA-BYW.10 (High Dose) Oral Vaccine — Enteric coated tablet for oral delivery
  Other Names: Influenza B (High Dose) Oral Vaccine Tablets
  Arms: VXA-BYW.10 (High Dose) Oral Vaccine
Other: Placebo Tablets — Enteric coated tablet for oral delivery
  Arms: Placebo Tablets

SUMMARY:
This is a phase 1, single-center, placeb-controlled, double-blind study. The purpose of this study is to determine the safety and immunogenicity of an oral vaccine tablet to prevent seasonal influenza B tested at two dose levels (low and high dose). The study will enroll 27 subjects in the low dose cohorts (3 sentinel open label subjects followed by 24 subjects (randomized 2:1 to vaccine vs placebo, respectively). Subsequently, 27 subjects will be enrolled in the high dose cohort in a similar manner as to the low dose cohort. Safety and immunogenicity will be evaluated at Day 28. Long term safety follow-up will be evaluated through 1 year post vaccination.

DETAILED DESCRIPTION:
The study will enroll 54 subjects in four cohorts. All subjects will receive a single administration of VXA-BYW.10 at a low dose, a high dose or placebo.

Two sentinel groups will enroll 3 subjects each in an open-label manner (Cohorts 1 and 3) to receive VXA-BYW.10 prior to enrolling either of the randomized, controlled cohorts (Cohorts 2 and 4). Within the double-blinded Cohorts (2 and 4), placebo subjects will receive the same number of tablets as the vaccine subjects in that Cohort. Subjects will be enrolled and dosed in the low dose groups prior to initiation of dosing in the high dose group.

Cohort 1: 3 subjects at low dose; Cohort 2: 16 subjects at low dose and 8 placebo; Cohort 3: 3 subjects at high dose; Cohort 4: 16 subjects at low dose and 8 placebo

Subjects will be followed for 28 days post vaccination for preliminary immunogenicity. Subjects will continue to be followed for 1 year post-vaccination for long term safety.

ELIGIBILITY:
Inclusion Criteria:

* In good health as established by medical history, physical examination, and laboratory testing at the time of enrollment.

Exclusion Criteria:

* Positive for B influenza by HAI.
* Has had an influenza vaccine in the past 2 years.
* Current history of chronic alcohol use and/or illicit and/or recreational drug use.
* History of any confirmed or suspected immunodeficient or immunosuppressive condition
* Positive serology for HIV, HCV, or HBV
* Previous serious reactions to vaccination such as anaphylaxis, respiratory problems, hives, or abdominal pain.
* History of irritable bowel disease or other inflammatory digestive or gastrointestinal conditions that could affect the intended distribution of the vaccine targeting the mucosa of the small intestine
* Use of proton pump inhibitors(Nexium, Prilosec).
* Stool sample with occult blood at baseline exam
* Pregnancy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Single High Dose of an Oral Influenza B Tablet Vaccine | Day 28
  Safety determined by reported solicited (reactogenicity) and unsolicited AEs.

SECONDARY OUTCOMES:
Immunogenicity of Single high Dose of an Oral Influenza B Tablet Vaccine | Day 28
  Efficacy determined by HAI titers at Day 28 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: David Liebowitz, MD, PhD, Study Director — Vaxart, Inc.
Locations (1):
- CCST, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No